CLINICAL TRIAL: NCT05404217
Title: A Randomized, Double-blind, Placebo-controlled Parallel-group Clinical Trial to Investigate the Efficacy and Safety of LN-OS-22 on Oxidative Stress and Systemic Inflammation in Overweight and Obese Population.
Brief Title: Clinical Trial to Investigate the Efficacy and Safety of LN-OS-22 on Oxidative Stress and Systemic Inflammation in Overweight and Obese Population.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: LI/211202/SOPH/OSSI
Record Dates: First submitted 2022-05-30; First posted 2022-06-03 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Oxidative Stress
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled parallel-group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LN-OS-22 (Active Comparator): 2 capsules orally once a day for 56 days
  Interventions: Other: LN-OS-22
- Maltodextrin (Placebo Comparator): 2 capsules orally once a day for 56 days
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: LN-OS-22 — 2 capsules orally once a day to be taken with a glass of milk after breakfast for 56 days
  Arms: LN-OS-22
Other: Maltodextrin — 2 capsules orally once a day to be taken with a glass of milk after breakfast for 56 days
  Arms: Maltodextrin

SUMMARY:
The present clinical investigation has been proposed to further substantiate the evidence of the antioxidant and anti-inflammatory activity of the extract in the healthy adult population with BMI ranging from ≥25.0 kg/m2 and ≤ 34.9 kg/m2 . The antioxidant effect of the 56 days of oral administration of the extract (1000 mg/day) will be primarily assessed by change in the level of 8-isoprostane from baseline to the end of the study and the anti-inflammatory activity of the extract will be investigated by the change in the level of CRP and IL-6. In addition, the effect on lipid peroxidation and DNA damage will be assessed by serum level of MDA before and after 2 months of extract administration. Further, metabolic endotoxemia will be assessed by the change in the plasma level of lipopolysaccharides. Weight and waist circumference are included as secondary outcomes as the clinical indicators of reduction in oxidative stress and inflammation. Overweight and obesity significantly impact the health-related quality of life31 in the affected individuals and flavonoids have previously been shown to improve the quality of life in controlled clinical studies therefore, Investigator included health-related quality of life as a secondary objective of the study. The safety of the 2-month administration of the extract will be examined by a change in the vitals, liver, and kidney function biomarkers (SGOT, SGPT, ALP, and creatinine).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥30 -≤60 years.
2. No history of systemic infection as assessed by normal total leucocyte count.
3. Overweight and obese participants (at high risk of oxidative stress and inflammation) identified as BMI ≥ 25.0 kg/m2 and ≤ 34.9 kg/m2
4. Individuals having a risk of metabolic syndrome as indicated by three or more of the following five criteria:

   a Waist circumference more than 102 cm for males or 88 cm for females b Blood pressure of more than 130/85 mmHg c Fasting triglyceride (TG) level ≥ 150 mg/dl d Fasting high-density lipoprotein cholesterol level ≤ 40 mg/dl for males or 50 mg/dl for females e Fasting blood glucose ≥ 100 mg/dl.
5. Individuals physically inactive for 1/3rd of the wake time as per the Longitudinal Aging Study Amsterdam (LASA) sedentary behavior questionnaire
6. Non-smokers (Past smokers can be allowed if they have abstinence for a minimum of 2 years)
7. Able to comply and perform the procedures requested by the protocol (including dietary restrictions, consumption of study interventions, blood and urine sample collection procedures, and study visit schedule)
8. Participants who are literate enough to read and understand the consent form and provide voluntary consent.
9. Participants who can give written informed consent and willing to participate in the study and comply with its procedures.

Exclusion Criteria:

1. Known sensitivity to the investigational product or any excipients of the drug product.
2. Known case of lactose intolerance.
3. Known case of type I diabetes.
4. Presence of uncontrolled type II diabetes mellitus (indicated by HbA1c ≥ 6.5).
5. Presence of uncontrolled hypertension (defined as Systolic Blood Pressure (SBP) ≥ 140 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 90 mm Hg).
6. Presence thyroid dysfunction (defined as thyroid stimulating hormone (TSH) level < 0.4 to > 4.2 mIU/L).
7. Participants with moderate to severe anemia defined as hemoglobin <10 gm/dL- in the case of females and < 11 gm/dL- in the case of males will be excluded from the study.
8. Consumption of any herbal preparation, supplements, nutritional therapy, etc. which is expected to reduce oxidative stress within 1 month prior to screening and throughout the study period.
9. History of any significant neurological and psychiatric condition which may affect the participation and inference of the study's endpoints.
10. History of use of anti-inflammatory therapies for any ailments within 7 days prior to randomization.
11. Participation in other clinical trials in the last 3 months prior to screening
12. Participants with substance abuse problems (within 2 years) defined as:

    a Use of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.)/Nicotine dependence.

    b High-risk drinking as defined by the consumption of 4 or more alcohol-containing beverages on any day or 8 or more alcohol-containing beverages per week for women and 5 or more alcohol-containing beverages on any day or 15 or more alcohol-containing beverages per week for men.
13. Participants who have a clinically significant disorder such as cardiovascular, endocrine, respiratory, gastrointestinal, hepatobiliary, kidney, urinary, hematological, immunity, neuropsychiatric, musculoskeletal, inflammatory, and/or tumors.
14. Females who are pregnant/planning to be pregnant/lactating or taking any oral contraceptives.
15. Any condition that could, in the opinion of the investigator, preclude the participant's ability to successfully and safely complete the study or that may confound study outcomes

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Oxidative stress | days 0, day 28, and day 56.
  To measure the oxidative stress 8-iso-PGF2α which is considered the best biomarker of oxidative stress will be assessed in the serum of the participants enrolled in the study. The blood sample will then be sent to the laboratory for analysis of serum levels of 8-iso-PGF2α by sandwich ELISA technique using GENLISATM ELISA kits. The normal reference range of 8-iso-PGF2α is 2-34 pg/ml (median).
  oxidative stress as assessed by change in serum levels of 8-isoprostane

SECONDARY OUTCOMES:
Systemic inflammation CRP and IL - 6 | days 0, day 28, and day 56.
  blood sample will then be sent to the laboratory for estimation of CRP by RHELAX-CRP slide test based on the principle of agglutination. Serum IL-6 will be estimated by using GENLISATM ELISA kits. The normal reference range of CRP is <10 mg/L and that of IL-6 is 0-50 pg/mL.
Metabolic endotoxemia | days 0, and day 56.
  The samples will be sent to the laboratory for the assessment of LPS by sandwich ELISA technique using GENLISATM ELISA kits. Reference range: Median (IQR) = 18.4 (8.6-56.8) μg/ml. Metabolic endotoxemia as assessed by change in plasma lipopolysaccharide levels post high-fat diet from baseline compared to placebo.
Body weight | days 0, day 28, and day 56.
  Participants will be weighed on a calibrated digital weighing scale (with minimal clothing and bare feet) on the screening visit, day 0, and monthly follow-up visits before taking breakfast. The body weight measurement will be taken twice, and if the difference between the two readings is greater than 1 kg, then a third measurement will be taken.
  Higher the body weight represents the worst scoring , lower the body weight represents best scoring
Waist circumference | days 0, day 28, and day 56.
  The waist circumference will be measured (in cm) at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest, using stretch-resistant tape. The measurement will be taken twice, and if the difference between the two readings is greater than 1 cm, then a third measurement will be taken.
  Higher the waist circumference represents the worst scoring , lower the body weight represents best scoring
Impact of Weight on Quality of Life-Lite-Clinical Trials | days 0, day 28, and day 56.
  Quality of life as assessed by change in the scores of Impact of Weight on Quality of Life-Lite-Clinical Trials Version from baseline. The higher the score, the greater will be impairment in quality of life.85

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shalini Srivastava, MD medicine, Study Director — Vedic Lifesciences Pvt. Ltd.
Locations (3):
- India (3):
  - Ayush Nursing Home, Mumbai, Maharashtra
  - Dr. Awate's Clinic, Mumbai, Maharashtra
  - Metabol-Lifestyle metabolic syndrome clinic, Mumbai, Maharashtra

IPD SHARING:
Plan to Share IPD: Undecided